CLINICAL TRIAL: NCT00852410
Title: The Hemostatic and Hemodynamic Effects of Adrenaline During Endoscopic Sinus Surgery: Randomized Clinical Trial
Brief Title: The Hemostatic and Hemodynamic Effects of Adrenaline During Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Dr. A. Moshaver, University Of Toronto
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0001-A
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Sinusitis
Keywords: Endoscopic sinus surgery
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% lidocaine with 1:100000 adrenaline (Active Comparator): high dose adrenaline
  Interventions: Drug: 1% lidocaine with 1:100,000 adrenaline
- 1% lidocaine with 1:200,000 adrenaline (Active Comparator): low dose
  Interventions: Drug: 1% lidocaine with 1:200,000 adrenaline

INTERVENTIONS:
Drug: 1% lidocaine with 1:100,000 adrenaline — high dose
  Arms: 1% lidocaine with 1:100000 adrenaline
Drug: 1% lidocaine with 1:200,000 adrenaline — 1% lidocaine with 1:200,000 adrenaline
  Arms: 1% lidocaine with 1:200,000 adrenaline

SUMMARY:
Obtaining adequate hemostasis is crucial during endoscopic sinus surgery. Submucosal injection of local anaesthetic containing adrenaline has frequently been used to improve surgical milieu. However, injection of adrenaline has potential side effects including tachycardia, hypertension as well as inducing arrhythmia. The aim of this randomized clinical trial is to assess the hemodynamic and hemostatic effects of two different concentrations of adrenaline in local anaesthetic used during endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* recurrent acute sinusitis, chronic sinusitis, or nasal polyposis

Exclusion Criteria:

* bleeding disorders, under age of 18, history of cardiac disease or on antihypertensive medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Reduction of Intraoperative bleeding | during surgery

SECONDARY OUTCOMES:
hemodynamic fluctuation | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ali Moshaver, MD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Moshaver A, Lin D, Pinto R, Witterick IJ. The hemostatic and hemodynamic effects of epinephrine during endoscopic sinus surgery: a randomized clinical trial. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):1005-9. doi: 10.1001/archoto.2009.144. PMID 19841339